CLINICAL TRIAL: NCT01332006
Title: Intra-bone Cord Blood Transplantation for Hematological Malignancies Lacking a HLA Suitable Donor
Brief Title: Intra-bone Cord Blood Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Domenico Russo, Director, Università degli Studi di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBMCB - BS study
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-bone injection (Experimental): Intra-bone transplantation of hematopoietic stem cells from cord blood
  Interventions: Procedure: Intrabone injection; Biological: Intra-bone cord blood hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: Intrabone injection — All adults patients with hematological malignancies, lacking a HLA matched donor fulfilling the inclusion criteria, will undergo to intrabone HSC infusion of CB.
  Other Names: Intrabone Transplant
Biological: Intra-bone cord blood hematopoietic stem cell transplantation
Biological: Intra-bone cord blood hematopoietic stem cell transplantation — Intra-bone injection of CB hematopoietic SCs after conditioning regimen
  Other Names: No other name

SUMMARY:
For the great majority of hematological malignancies, hemopoietic stem cell (HSC) transplant is the only possible cure. The source of HSC is usually bone marrow (BM) or peripheral blood cell (PBSC) mobilized by granulocyte growth factor. Transplant needs a HLA compatible donor weather related or unrelated. A suitable compatible donor can be found in at least 70% of the patients. Thus, at least 30% of patients with indication for allogeneic HSC transplant are not able to undergo the procedure because of the lack of a HLA compatible donor. Cord blood (CB) cells represent another possible source, that needs a lower degree of HLA compatibility. CB transplant, however, offers a lower number of HSC. Thus, adult patient rarely may benefit from this source of stem cells, mainly beacuse thie body weight is too high to have ad adequate number of cell per kg. Recently, experimental animal models confirmed that an adequate recovery of allogeneic hemopoiesis can be achieved via intrabone injection, using a 1Log lower number of cells compared to the intravenous way (Yahata 2003, Castello 2004). Safety and feasibility of intrabone infusion was verified by two clinical studies on humans: the first was conducted by Ringden O. et al. in 18 patients using BM as a source of SC. No side effects and complete engraftment of donor hemopoiesis was observed; the second one was conducted by Frassoni et al. (Frassoni 2008) with CB as the source of HSC.

The aim of this study is to evaluate the intrabone infusion of compatible CB in patients with haematological malignancies lacking a HLA matched donor.

We will perform:

evaluation of the engraftment kinetics; evaluation of the chimerism degree at 30, 60, 100 days, 6 months and 1 year after transplant; studies on immunological reconstitution and the role of the NK compartment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Patients affected by hematological malignancies without a HLA identical sibling donor or unrelated donor.
* Informed consent.

Exclusion Criteria:

* Patients with ECOG < 2.
* Patients with blood creatine > 2 mg/dl or with transaminase or cholestase index > 5 times compared to normality upper limits.
* Patients with Cardiac Fraction Ejection < 40%.
* Patients with DLCO < 60% or Diffusing Lung Capacity of carbon monoxide attesting a severe pulmonary insufficiency.
* Patients with peripheral blast cell count over 10%.
* Second neoplasia diagnosed no more than 2 years before.
* Patients with active or suspected infection by fungi for which a therapeutic treatment is ongoing.
* HIV positive patients.
* HCV-RNA and HBV-DNA positive patients
* Pregnant or lactating women.
* Severe mental diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2009-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of transplanted patients with successful engraftment at day +30 | 30 days post transplantation
  Engraftment

SECONDARY OUTCOMES:
Clinical response with the analysis of global survival, survival without relapse, relapse incidence | 3 years from transplantation
Infections' Incidence | One year after transplantation
Chimerism monitoring on selected cell populations | Every three months and until one year after transplantation
Immunological reconstitution | One year after transplantation
Acute an Chronic GVHD | One year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Russo, Full Professor, Principal Investigator — USD TMO Adulti
Locations (1):
- USD TMO Adulti, Piazzale Spedali Civili, Brescia, Italy